CLINICAL TRIAL: NCT04672694
Title: Randomized Controlled Study of Effects of Intraoperative Vagal Block on Reducing the Postoperative Cough After Thoracic Surgery
Brief Title: Effects of Intraoperative Vagal Block on Reducing the Postoperative Cough After Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Seong Yong Park, Associate Professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2020-1087
Record Dates: First submitted 2020-12-06; First posted 2020-12-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Cough; Thoracic Surgery; Nerve Block
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNB (vagus nerve block) (Active Comparator): Vagus nerve block
  Interventions: Procedure: Vagus nerve block
- Control (Placebo Comparator): No vagus nerve block
  Interventions: Procedure: No vagus nerve block

INTERVENTIONS:
Procedure: Vagus nerve block — Ropivacine 0.75% 2mL will be injected two times around the vagus nerve (just below the bifurcation of recurrent laryngeal nerve); one before starting the surgical resection of lung including complete mediasitnal lymph node dissection and one at the end of operation.
  Arms: VNB (vagus nerve block)
Procedure: No vagus nerve block — No vagus nerve block will be conducted during the surgery.
  Arms: Control

SUMMARY:
Randomized controlled study to investigate the role of intraoperative vagal nerve block for preventing the postoperative cough in patients who received the pulmonary resection for lung cancer

DETAILED DESCRIPTION:
The standard treatments for early primary lung cancer are surgical treatments (lobectomy and lymph node resection). The usual mortality rate of lung cancer surgery is 1-2%, and the incidence of complications is reported to be about 20%. In addition to these deaths and complications, there are frequent sequelae such as reduction of pulmonary function reduction and cough. According to a cross section study of 240 patients who underwent lung cancer surgery, about 30% of patients complained of cough after surgery for one year after surgery, and 50% of patients complained of cough after one year. After the pulmonary resection of lung cancer, chronic coughs are the main cause of lowering the quality of life of patients after lung surgery. Several studies have reported the risk factors of cough after lung cancer surgery, and it is known that there is a relationship between mediastinal lymph node resection and accompanying gastric-esophageal gastric acid reflux.

According to anatomy and physiology studies of coughs, coughing occurs due to stimulation of vagus nerves, which is a type of reflex to protect the respiratory tract from harmful stimuli from the outside. Cough cough is known to occur when c-fibers are stimulated, especially at the end of the vagus nerve. Cough reflex-related circuits from c-fiber to brain are generated, and then coughing is reported in smaller stimuli. The end of the vagus nerves in the bronchial area can be damaged by the mediastinal lymph nodes dissection during lung cancer surgery and it can lead to c-fiber stimulation and finally form the nerve circuit which can lead to chronic cough.

Recently, awake pulmonary resection (awakening surgery) has been performed in several countries. Normally, sleep anesthesia gas itself is depleted of vagus nerve function and does not cause cough reflex during surgery, but when operated in a waking state, coughing caused by vagus nerve stimulation may occur and dangerous situations may occur during surgery, so it is reported that vagus nerve block is performed at the start of surgery. These vagus nerve blocks are known to prevent cough reflex during awakening surgery and enable surgery to be performed stably. However, it is not yet known whether these vagus nerve block can reduce acute and chronic cough after surgery. In this study, we investigated whether vagus nerve block during surgery could reduce coughing after surgery in patients who underwent general anesthesia lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' physical status class Ⅲ
* Diagnosed with non-small cell lung cancer with clinical stage of I-IIIA
* Planned to undergo segmentectomy or lobectomy with mediastinal lymph node dissection

Exclusion Criteria:

* chronic cough symptoms before surgery; a chronic cough (a cough lasting more than eight weeks)
* chemotherapy or chemoradiotherapy prior to surgery
* current smoker (patient should quit smoking at least 2 weeks before surgery)
* previously diagnosed with airway disease prior to surgery
* previously diagnosed with asthma prior to surgery
* patients with nervous system defects or psychiatric problems
* patients with severe cardiovascular disease, hepatological, or renal failure

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Cough score | 6 months after surgery
  The cough score is a two-part questionnaire referring to a symptoms during the day and night time. The response scale captures cough frequency, intensity and overall impact.

SECONDARY OUTCOMES:
COAT, Cough Assessment Test | 6 months after surgery
  The COAT is a short, simple questionnaire that assesses cough frequency, limitation on daily activities, sleep disturbance, fatigue and hypersensitivity to irritants in recent 1 week. It consists of five items, each with a 5-point differential scale (0-4), constituting a 0-20-point total scale.
Cough numeric rating scales (NRS) | 6 months after surgery
  The cough NRS range from 0 (no cough at all) to 10 (maximal cough).
Leicester cough questionnaire | 6 months after surgery
  LCQ is a validated self-reporting quality of life measures of cough in recent 2 weeks. It consists of 19 items with a 7 point likert response scale (range from 1 to 7) and it takes less than 5 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Yong Park, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No